CLINICAL TRIAL: NCT05789277
Title: Effects of Eccentric Hamstring Training, in Prevention of Hamstring Injuries in Sports Involving Sprinting Among Club Level Athletes
Brief Title: Effects of Eccentric Hamstring Training in Prevention of Hamstring Injuries in Sprinters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/01407 MOHAIB JONATHAN
Record Dates: First submitted 2023-02-28; First posted 2023-03-29 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-04

CONDITIONS: Sport Injury
Keywords: athletic injuries; hamstring; eccentric training; prevention; sprinters
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional training program group (Active Comparator): The control group will perform conventional training program
  Interventions: Other: Conventional training program
- Eccentric hamstring training group (Experimental): The interventional group will perform eccentric hamstring training
  Interventions: Other: Eccentric hamstring training

INTERVENTIONS:
Other: Conventional training program — Conventional training program:
  5-10 Repetitions ( 0.5-to 1-min rest);
  1. Vertical jumps
  2. Multiple forward jumps
  3. Running exercises
  4. Sprints alternating with slow jogging
  Arms: Conventional training program group
Other: Eccentric hamstring training — Functional training along with specific eccentric hamstrings exercises i.e., prone hamstring curl, exercise ball (or glider) bridge with curl, Nordic hamstring curl, single leg deadlift. The exercise program comprises 3 sets of 15 repetitions once to twice per day for at least 12 weeks.
  Arms: Eccentric hamstring training group

SUMMARY:
The goal of this clinical trail is to determine the effects of eccentric hamstring training, in prevention of hamstring injuries in sports involving sprinting among club level athletes.

The main question it aims to answer is :

- Will eccentric exercises have an effect in the recovery of hamstring injuries and injury prevention in sprint performance sports among club-level athletes.

Participants will be divided into two groups. Control group will perform conventional training program and interventional group will perform eccentric exercises.

DETAILED DESCRIPTION:
The most frequent time-loss injuries in sports are hamstring injuries, which are particularly common in modalities that involve rapid accelerations and decelerations like high-speed running. The hamstring muscle group is more susceptible to stresses because of the way it is anatomically arranged.These injuries are more common in sprinters than in other athletes.Ballistic motions like sprinting are typical in most contact and non-contact sports. The most frequent type of activity during sprinting is the running stride. The muscles aggressively extend and contract throughout each stride, forcing the linked segments to accelerate and slow down.In most club-level sports like football, cricket, sprinters and rugby sprinting is a crucial component of the sports and defines the performance of the athletes. If the athlete is a good sprinter he will perform more efficiently in sports. As sprinting is a high-intensity activity and is beneficial for athlete's general health but there are many injuries involved among these athletes. The injury can be disastrous for the athlete, resulting in extended recovery time and the possibility of persistent damage. Injuries in professional athletes are disproportionately often hamstring-related.The most common form of hamstring injury is hamstring strain which can be caused due these reasons. Hamstring injuries can be divided into three types; Grade 1 which is a hamstring pull or strain, Grade 2 partial muscle tear and Grade 3 complete muscle tear. The hamstring muscle is very important as it is involved in generating forward motion. The cause of hamstring injury can be due to multiple activities but the most common is when athletes are sprinting at maximal speeds.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 28 years.
* Rugby players
* Male
* Athletes who have suffered a hamstring injury in the past 6 months.

Exclusion Criteria:

* Those athletes who have undergone any surgery in the lower extremity and athletes with any other lower limb pathology are excluded.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Functional Assessment Scale for acute hamstring injury | The participants will be assessed at Baseline, 4th week, 12th week and 24th week
  FASH (Functional Assessment Scale for Acute Hamstring Injuries) questionnaire has recently been developed as a disease-specific and self-administered questionnaire to grade the severity of symptoms (pain and function) in patients with hamstring injuries.
  The FASH consists of six items, each of which is scored on a scale of 0 to 10, with 0 indicating the worst possible function and 10 indicating the normal function. The total score on the FASH ranges from 0 to 60, with higher scores indicating better function.
Change in Nordic Hamstring Exercise test: | The participants will be assessed at Baseline, 4th week, 12th week and 24th week
  The nordic hamstring exercise test is used to determine the effectiveness of the Nordic hamstring exercise program on Nordic hamstring exercise performance. From a kneeling position on the device, with the ankles secured under a heavy lifting sling, participants leaned forward in a controlled manner as far as possible (eccentric phase) and then returned to the starting position (concentric phase). A tape measure documented the forward distance achieved by the participants in cm.
Change in Single Leg Hamstring Bridge test | The participants will be assessed at Baseline, 4th week, 12th week and 24th week
  A single-leg hamstring bridge to assess the functional strength of the hamstring muscle group. This activity is performed with the injured limb propped on a 60 cm surface at 20oknee flexion, (plyo box, chair, exercise ball) while the unaffected limb is held in the air. The pelvis is then lifted off the ground in the motion of a bridge. This places demand directly on the hamstring to contract to support the body during the bridge.
Change in Lasegue (Straight leg raise test): | The participants will be assessed at Baseline, 4th week, 12th week and 24th week
  The straight leg raise test measures hamstring tightness. Restricted flexibility in the hamstrings will contribute to lower back, pelvis, hip, and knee mal-alignment. The straight leg raise test focuses on proximal hamstring tightness. The test is performed passively.
Change in Slump test with cervical flexion & extension: | The participants will be assessed at Baseline, 4th week, 12th week and 24th week
  Addressing the lumbar spine and pelvic joints may be important as the presence of pain referred into the leg can change hamstring strength, muscle contraction timing, and willingness to bend. Manual pain provocation tests may be used to clear the lumbopelvic region in the hamstring-injured patient, and the slump test may be used to differentiate hamstrings and sciatic nerve symptoms as the source of posterior thigh pain.The slump test is positive where the patient's posterior thigh pain is reproduced in the final slump position, and reduced with cervical extension.
Change in 20m Multistage Fitness Test (Beep Test) | The participants will be assessed at Baseline, 4th week, 12th week and 24th week
  The 20m multistage fitness test (MSFT) also known as 20 meter shuttle run test or beep test is a commonly used maximal running aerobic fitness test. The equipment required for this test are flat, non-slip surface, marking cones, 20m measuring tape,beep test audio, audio player, recording sheets.This test involves continuous running between two lines 20m apart in time to recorded beeps. The participants start running when the recording tells them to,standing behind one line and facing the other. The first speed is really slow. The subject keeps moving between the two lines while turning when the beeps are captured. The beeps will get more frequent and louder after about a minute, and a sound will signal an increase in speed.The level and number of shuttles (20m) the athlete completed before they were unable to keep up with the recording determines their score.

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Rugby Ground, Sector F-10/1, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No